CLINICAL TRIAL: NCT01065454
Title: Randomized, Double Blind, Placebo Controlled, Parallel Group, Multi-center Study to Evaluate the Hemodynamic Effects of Riociguat (BAY 63-2521) as Well as Safety and Kinetics in Patients With Pulmonary Hypertension Associated With Left Ventricular Systolic Dysfunction
Brief Title: A Study to Test the Effects of Riociguat in Patients With Pulmonary Hypertension Associated With Left Ventricular Systolic Dysfunction
Acronym: LEPHT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14308; 2023-507001-34-00 (Other: CTIS (EU)); 2009-015878-35 (EudraCT Number)
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Results first posted 2013-12-25 (Estimated); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Hypertension, Pulmonary; Ventricular Dysfunction, Left
Keywords: Pulmonary Hypertension; Left ventricular dysfunction
MeSH Terms: conditions — Hypertension, Pulmonary; Ventricular Dysfunction, Left | interventions — riociguat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Riociguat (Adempas, BAY63-2521) up to 2 mg (Experimental): Participants received riociguat up to 2 mg three times per day (tid) (increasing from 0.5 to 1 to 2 mg).
  Interventions: Drug: Riociguat (Adempas, BAY63-2521)
- Riociguat (Adempas, BAY63-2521) up to 1 mg (Experimental): Participants received riociguat up to 1 mg tid (increasing from 0.5 to 1 mg).
  Interventions: Drug: Riociguat (Adempas, BAY63-2521)
- Riociguat (Adempas, BAY63-2521) fixed 0.5 mg (Experimental): Participants received riociguat 0.5 mg tid (fixed dose).
  Interventions: Drug: Riociguat (Adempas, BAY63-2521)
- Placebo (Placebo Comparator): Participants received placebo tid.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Riociguat (Adempas, BAY63-2521) — up to 2 mg three times a day (increasing from 0.5 to 1 to 2 mg)
  Arms: Riociguat (Adempas, BAY63-2521) up to 2 mg
Drug: Riociguat (Adempas, BAY63-2521) — up to 1 mg three times a day (increasing from 0.5 to 1 mg)
  Arms: Riociguat (Adempas, BAY63-2521) up to 1 mg
Drug: Riociguat (Adempas, BAY63-2521) — fixed 0.5 mg three times a day
  Arms: Riociguat (Adempas, BAY63-2521) fixed 0.5 mg
Drug: Placebo — Placebo three times a day
  Arms: Placebo

SUMMARY:
The aim of this study is to assess whether increasing oral doses of Riociguat are safe and improve the well-being, symptoms and outcome in patients with pulmonary hypertension associated with left ventricular systolic dysfunction

DETAILED DESCRIPTION:
Pharmacokinetics parameters were regarded as exploratory parameters. Adverse event data will be covered in Adverse events section.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with symptomatic pulmonary hypertension due to left ventricular systolic dysfunction despite optimized heart failure therapy

Exclusion Criteria:

* Types of pulmonary hypertension other than group 2.1 of Dana Point Classification

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2010-04-14 (Actual); Primary Completion 2012-06-06 (Actual); Study Completion 2025-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (78):
- United States (14):
  - Los Angeles, California
  - San Diego, California
  - Torrance, California
  - Westminster, California
  - Miami, Florida
  - Iowa City, Iowa
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Rochester, Minnesota
  - St Louis, Missouri
  - Cincinnati, Ohio
  - Fairfield, Ohio
  - Falls Church, Virginia
  - Milwaukee, Wisconsin
- Australia (3):
  - Sydney, New South Wales
  - Herston, Queensland
  - Melbourne, Victoria
- Austria (2):
  - Innsbruck, Tyrol
  - Vienna
- Belgium (4):
  - Aalst
  - Brussels
  - Ghent
  - Leuven
- Canada (4):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Montreal, Quebec
  - Québec
- China (2):
  - Beijing
  - Shanghai
- Czechia (3):
  - Brno
  - Olomouc
  - Prague
- Aarhus N, Denmark
- France (6):
  - Bron
  - Lille
  - Nantes
  - Pessac
  - Rouen
  - Toulouse
- Germany (5):
  - Heidelberg, Baden-Wurttemberg
  - Augsburg, Bavaria
  - Greifswald, Mecklenburg-Vorpommern
  - Cologne, North Rhine-Westphalia
  - Erfurt, Thuringia
- Italy (2):
  - Naples, Campania
  - Pavia, Lombardy
- Japan (14):
  - Nagoya, Aichi-ken
  - Seto, Aichi-ken
  - Ōgaki, Gifu
  - Higashiibaraki, Ibaraki
  - Tsu, Mie-ken
  - Sendai, Miyagi
  - Kita-ku, Osaka, Osaka
  - Osaka, Osaka
  - Suita, Osaka
  - Kusatsu, Shiga
  - Sunto, Shizuoka
  - Arakawa-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Tanabe, Wakayama
- Netherlands (2):
  - Amsterdam
  - Nijmegen
- Poland (3):
  - Bydgoszcz
  - Gdansk
  - Warsaw
- Singapore, Singapore
- Spain (7):
  - A Coruña, A Coruña
  - Majadahonda, Madrid
  - Palma, Palma de Mallorca
  - Barcelona
  - Madrid
  - Murcia
  - Valencia
- Switzerland (3):
  - Geneva, Canton of Geneva
  - Lugano, Canton Ticino
  - Zurich
- United Kingdom (2):
  - Cambridge, Cambridgeshire
  - London

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Result] Ghio S, Bonderman D, Felix SB, Ghofrani HA, Michelakis ED, Mitrovic V, Oudiz RJ, Frey R, Roessig L, Semigran MJ. Left ventricular systolic dysfunction associated with pulmonary hypertension riociguat trial (LEPHT): rationale and design. Eur J Heart Fail. 2012 Aug;14(8):946-53. doi: 10.1093/eurjhf/hfs071. Epub 2012 Jun 20. PMID 22719060
- [Result] Bonderman D, Ghio S, Felix SB, Ghofrani HA, Michelakis E, Mitrovic V, Oudiz RJ, Boateng F, Scalise AV, Roessig L, Semigran MJ; Left Ventricular Systolic Dysfunction Associated With Pulmonary Hypertension Riociguat Trial (LEPHT) Study Group. Riociguat for patients with pulmonary hypertension caused by systolic left ventricular dysfunction: a phase IIb double-blind, randomized, placebo-controlled, dose-ranging hemodynamic study. Circulation. 2013 Jul 30;128(5):502-11. doi: 10.1161/CIRCULATIONAHA.113.001458. Epub 2013 Jun 17. PMID 23775260

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only subjects with symptomatic pulmonary hypertension associated with left ventricular systolic dysfunction (PH-sLVD) could participate in this study. Subjects must have been pre-treated with optimized CHF therapy.
Pre-assignment Details: 301 subjects were screened in 84 study centers in 18 countries worldwide. 99 of the 301 screened subjects were not randomized (adverse event [1], protocol violation [1], screen failure [87], withdrawal by subject [10]). Of the 202 subjects randomized, one subject did not receive any study medication.
Period: Treatment
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2 mg | Riociguat (Adempas, BAY63-2521) up to 1 mg | Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg | Placebo
Started | 67 | 33 | 32 | 69
Completed | 54 | 28 | 23 | 57
Not Completed | 13 | 5 | 9 | 12
Not completed — Adverse Event | 7 | 4 | 3 | 6
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Non-compliance | 1 | 0 | 0 | 1
Not completed — Protocol Decision | 0 | 0 | 3 | 2
Not completed — Protocol Violation | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 2 | 3
Period: Follow up
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2 mg | Riociguat (Adempas, BAY63-2521) up to 1 mg | Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg | Placebo
Started | 54 | 28 | 23 | 57
Entering Follow-up | 49 | 27 | 23 | 51
Completed | 15 | 4 | 6 | 13
Not Completed | 39 | 24 | 17 | 44
Not completed — Adverse Event | 1 | 0 | 0 | 1
Not completed — Death | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Progressive disease | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0
Not completed — study ongoing | 37 | 22 | 15 | 41

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2 mg | Riociguat (Adempas, BAY63-2521) up to 1 mg | Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg | Placebo | Total
Number analyzed (Participants) | 67 | 33 | 32 | 69 | 201
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.3 (10.8) | 55.1 (13.2) | 57.2 (9.9) | 58.9 (11.2) | 58.1 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 3 | 6 | 8 | 29
  Male | 55 | 30 | 26 | 61 | 172
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 28.87 (5.27) | 28.16 (4.72) | 29.20 (5.64) | 28.65 (5.89) | 28.73 (5.44)
6-minute walking distance [Mean (Standard Deviation); unit: Meters] — 6MWD is a measure for the evaluation of functional exercise capacity.
  Meters | 380.9 (125.80) | 401.9 (101.75) | 416.6 (95.77) | 382.1 (123.51) | 390.5 (116.94)
Left ventricular ejection fraction (LVEF) [Mean (Standard Deviation); unit: Percentage] — LVEF is a calculated echocardiography parameter.
  Percentage | 28.4 (5.72) | 28.8 (4.54) | 27.0 (5.21) | 27.1 (5.02) | 27.8 (5.24)
Etiology [Count of Participants; unit: Participants]
  Ischemic cardiomyopathy | 30 | 12 | 14 | 34 | 90
  Non-ischemic cardiomyopathy | 37 | 20 | 17 | 34 | 108
  Data missing | 0 | 1 | 1 | 1 | 3
WHO (World Health Organization) functional class [Count of Participants; unit: Participants] — The WHO functional assessment of pulmonary arterial hypertension ranged from functional class I (Patients with PH but without resulting limitation of physical activity) to class IV (Patients with PH with inability to carry out any physical activity without symptoms. These patients manifest signs of right-heart failure.). Changes to a lower WHO functional class resemble improvement, changes to a higher functional class resemble deterioration of pulmonary arterial hypertension (PAH).
  Participants
    II | 35 | 20 | 23 | 42 | 120
    III | 31 | 13 | 9 | 23 | 76
    IV | 1 | 0 | 0 | 4 | 5
Number of participants with diabetes mellitus (including subtypes) [Count of Participants; unit: Participants] | 30 | 10 | 13 | 34 | 87
Glomerular filtration rate (GFR) [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 65.1 (19.10) | 72.6 (22.70) | 72.0 (17.90) | 68.7 (19.90) | 68.7 (19.91)
Number of participants with atrial fibrillation [Count of Participants; unit: Participants] | 9 | 3 | 3 | 9 | 24
Number of participants with atrial flutter [Count of Participants; unit: Participants] | 0 | 0 | 1 | 1 | 2
Number of participants with pacemaker rhythm [Count of Participants; unit: Participants] | 17 | 9 | 7 | 17 | 50
Baseline drug and device therapy [Count of Participants; unit: Participants] — A single patient could have more than one drug and device therapy.
  Participants
    Cardiac devices | 38 | 17 | 21 | 44 | 120
    Angiotensin-converting enzyme inhibitors | 50 | 25 | 21 | 46 | 142
    Angiotensin II receptor blockers | 20 | 8 | 10 | 19 | 57
    Aldosterone antagonists | 51 | 26 | 23 | 53 | 153
    Beta-blockers | 31 | 16 | 21 | 32 | 100
    Beta-blockers with alpha-blocking activity | 30 | 15 | 11 | 30 | 86
    Loop diuretics | 62 | 31 | 29 | 68 | 190
    Thiazide diuretics | 12 | 3 | 7 | 10 | 32
    Cardiac glycosides | 28 | 12 | 6 | 28 | 74
    Oral anticoagulants | 38 | 16 | 15 | 33 | 102
    Amiodarone | 9 | 3 | 4 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Pulmonary Artery Mean Pressure (PAPmean) at Rest - Change From Baseline to Week 16
Description: Mean pulmonary arterial pressure (PAPmean) is a directly measured hemodynamic parameter. PAPmean is recorded during a right heart catheterization.
Time Frame: Baseline and visit 6 (16 weeks)
Population: Per-protocol set (PPS) - A subject was included in the PPS if he/she was valid for SAF [safety analysis set]/ITT and showed no major protocol deviations affecting efficacy. Only participants with a baseline and at least one post-baseline measurement were included in this analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2 mg | Riociguat (Adempas, BAY63-2521) up to 1 mg | Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg | Placebo
Number analyzed (Participants) | 54 | 28 | 22 | 56
mmHg | -6.1 (9.68) | -0.8 (8.41) | -4.5 (7.35) | -4.0 (9.00)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) up to 2 mg vs Placebo; Test type: Superiority or Other; p = 0.1044, ANCOVA — Baseline value, treatment group and region were used as fixed effects in the ANCOVA model; LS-MEANS Difference = -2.71, 95% CI 2-sided [-5.99 to 0.057]
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521) up to 2 mg vs Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg; Test type: Superiority or Other; p = 0.5292, ANCOVA — Baseline value, treatment group and region were used as fixed effects in the ANCOVA model; LSMEANS Difference = -1.38, 95% CI 2-sided [-5.71 to 2.94]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521) up to 2 mg vs Riociguat (Adempas, BAY63-2521) up to 1 mg; Test type: Superiority or Other; p = 0.0278, ANCOVA — Baseline value, treatment group and region were used as fixed effects in the ANCOVA model; LS-MEANS Difference = -4.51, 95% CI 2-sided [-8.52 to -0.50]
Statistical Analysis 4: Comparison: Riociguat (Adempas, BAY63-2521) up to 1 mg vs Placebo; Test type: Superiority or Other; p = 0.3821, ANCOVA — Baseline value, treatment group and region were used as fixed effects in the ANCOVA model; LS-MEANS Difference = 1.80, 95% CI 2-sided [-2.25 to 5.84]
Statistical Analysis 5: Comparison: Riociguat (Adempas, BAY63-2521) up to 1 mg vs Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg; Test type: Superiority or Other; p = 0.2084, ANCOVA — Baseline value, treatment group and region were used as fixed effects in the ANCOVA model; LS-MEANS Difference = 3.13, 95% CI 2-sided [-1.76 to 8.02]
Statistical Analysis 6: Comparison: Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg vs Placebo; Test type: Superiority or Other; p = 0.5442, ANCOVA — Baseline value, treatment group and region were used as fixed effects in the ANCOVA model; LS-MEANS Difference = -1.33, 95% CI 2-sided [-5.66 to 3.00]

2. Secondary Outcome: Venous Oxygen Saturation (SvO2) - Change From Baseline to Week 16
Description: The mixed venous oxygen saturation rate (SvO2) is a directly measured hemodynamic parameter. SvO2 is recorded during a right heart catheterization.
Time Frame: Baseline and visit 6 (16 weeks)
Population: Per-protocol set (PPS) - A subject was included in the PPS if he/she was valid for SAF/ITT and showed no major protocol deviations affecting efficacy. Only participants with a baseline and at least one post-baseline measurement were included in this analysis.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2 mg | Riociguat (Adempas, BAY63-2521) up to 1 mg | Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg | Placebo
Number analyzed (Participants) | 45 | 23 | 19 | 48
Percentage | 1.98 (7.084) | 0.46 (7.866) | -0.21 (5.969) | 1.28 (9.259)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) up to 2 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = 1.87, 95% CI 2-sided [-0.83 to 4.56]
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521) up to 1 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = 0.20, 95% CI 2-sided [-3.12 to 3.51]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = 0.23, 95% CI 2-sided [-3.31 to 3.77]

3. Secondary Outcome: Pulmonary Vascular Resistance (PVR) - Change From Baseline to Week 16
Description: The pulmonary vascular resistance (PVR) is a calculated hemodynamic parameter. PVR is derived from the directly measured parameters mean pulmonary arterial pressure (PAPmean) and pulmonary capillary wedge pressure (PCWP), divided by the cardiac output (CO). PVR and PAPmean are acquired during a right heart catheterization. CO is a calculated hemodynamic parameter, too. Formula: PVR = 80*(PAPmean - PCWP)/CO
Time Frame: Baseline and visit 6 (16 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: dyn*s*cm^-5
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2 mg | Riociguat (Adempas, BAY63-2521) up to 1 mg | Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg | Placebo
Number analyzed (Participants) | 53 | 28 | 22 | 56
dyn*s*cm^-5 | -78.15 (125.261) | -33.05 (99.322) | -51.44 (124.107) | -36.97 (157.523)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) up to 2 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -46.59, 95% CI 2-sided [-89.4 to -3.8]
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521) up to 1 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -32.26, 95% CI 2-sided [-84.9 to 20.4]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -26.52, 95% CI 2-sided [-83.0 to 30.0]

4. Secondary Outcome: Pulmonary Vascular Resistance Index (PVRi) - Change From Baseline to Week 16
Description: The pulmonary vascular resistance index (PVRi) is a calculated hemodynamic parameter. PVRi is derived from the pulmonary vascular resistance (PVR) normalized by the body surface area (BSA). Formula: PVRi = 80*(PAPmean - PCWP)*BSA/CO
Time Frame: Baseline and visit 6 (16 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: dyn*s*cm^-5*m^2
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2 mg | Riociguat (Adempas, BAY63-2521) up to 1 mg | Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg | Placebo
Number analyzed (Participants) | 53 | 27 | 22 | 56
dyn*s*cm^-5*m^2 | -152.60 (250.366) | -61.763 (202.138) | -91.65 (237.256) | -76.47 (311.693)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) up to 2 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -89.17, 95% CI 2-sided [-172.9 to 5.5]
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521) up to 1 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -58.22, 95% CI 2-sided [-162.1 to 45.6]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -43.22, 95% CI 2-sided [-153.7 to 67.1]

5. Secondary Outcome: Systemic Vascular Resistance (SVR) - Change From Baseline to Week 16
Description: The systemic vascular resistance (SVR) is a calculated hemodynamic parameter. SVR is derived from the directly measured parameter mean right atrial pressure (RAPmean) and the calculated parameter mean systemic arterial pressure (SAPmean) divided by the cardiac output (CO). RAPmean is acquired during a right heart catheterization. CO is a calculated hemodynamic parameter, too. Formula: SVR = 80*(SAPmean - RAPmean)/CO
Time Frame: Baseline and visit 6 (16 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: dyn*s*cm^-5
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2 mg | Riociguat (Adempas, BAY63-2521) up to 1 mg | Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg | Placebo
Number analyzed (Participants) | 53 | 27 | 22 | 56
dyn*s*cm^-5 | -340.44 (394.87) | -118.72 (369.865) | -67.46 (315.097) | -94.37 (431.049)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) up to 2 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -239.31, 95% CI 2-sided [-363.4 to -115.3]
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521) up to 1 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -120.89, 95% CI 2-sided [-274.4 to 32.6]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -25.54, 95% CI 2-sided [-189.3 to 138.2]

6. Secondary Outcome: Systemic Vascular Resistance Index (SVRi) - Change From Baseline to Week 16
Description: The systemic vascular resistance index (SVRi) is a calculated hemodynamic parameter. SVRi is derived from the systemic vascular resistance (SVR) normalized by the body surface area (BSA). Formula: SVRi = 80*(SAPmean - RAPmean)*BSA/CO
Time Frame: Baseline and visit 6 (16 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: dyn*s*cm^-5*m^2
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2 mg | Riociguat (Adempas, BAY63-2521) up to 1 mg | Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg | Placebo
Number analyzed (Participants) | 53 | 27 | 22 | 56
dyn*s*cm^-5*m^2 | -651.98 (757.617) | -217.14 (742.465) | -100.31 (612.460) | -195.11 (853.927)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) up to 2 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -446.49, 95% CI 2-sided [-687.4 to -205.6]
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521) up to 1 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -231.57, 95% CI 2-sided [-530.4 to 67.2]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -34.97, 95% CI 2-sided [-353.7 to 283.7]

7. Secondary Outcome: Transpulmonary Pressure Gradient (TPG) - Change From Baseline to Week 16
Description: The transpulmonary pressure gradient (TPG) is a calculated hemodynamic parameter. TPG is calculated from the directly measured parameters mean pulmonary arterial pressure (PAPmean) and pulmonary capillary wedge pressure (PCWP). These 2 parameters are acquired during a right heart catheterization. Formula: TPG = PAPmean - PCWP
Time Frame: Baseline and visit 6 (16 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2 mg | Riociguat (Adempas, BAY63-2521) up to 1 mg | Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg | Placebo
Number analyzed (Participants) | 53 | 28 | 22 | 56
mmHg | -2.16 (4.795) | -1.01 (5.224) | -1.65 (4.652) | -1.37 (7.001)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) up to 2 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -1.27, 95% CI 2-sided [-3.1 to 0.5]
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521) up to 1 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -0.88, 95% CI 2-sided [-3.1 to 1.3]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -0.84, 95% CI 2-sided [-3.2 to 1.5]

8. Secondary Outcome: Pulmonary Capillary Wedge Pressure (PCWP) - Change From Baseline to Week 16
Description: Pulmonary capillary wedge pressure (PCWP) is a directly measured hemodynamic parameter acquired during a right heart catheterization.
Time Frame: Baseline and visit 6 (16 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2 mg | Riociguat (Adempas, BAY63-2521) up to 1 mg | Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg | Placebo
Number analyzed (Participants) | 53 | 28 | 22 | 56
mmHg | -3.93 (9.381) | 0.25 (9.001) | -2.818 (7.842) | -2.68 (7.791)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) up to 2 mg vs Placebo; Test type: Superiority or Other; LSS-MEANS Difference = -2.07, 95% CI 2-sided [-5.0 to 0.8]
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521) up to 1 mg vs Placebo; Test type: Superiority or Other; Ls Means = 1.39, 95% CI 2-sided [-2.1 to 4.9]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg vs Placebo; Test type: Superiority or Other; LS_MEANS Difference = -1.13, 95% CI 2-sided [-4.9 to 2.7]

9. Secondary Outcome: Tricuspid Annular Plane Systolic Excursion (TAPSE) - Change From Baseline to Week 16
Description: The tricuspid annular plane systolic excursion (TAPSE) is a measured echocardiography parameter. It is acquired during a non-invasive echocardiography examination.
Time Frame: Baseline and visit 6 (16 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2 mg | Riociguat (Adempas, BAY63-2521) up to 1 mg | Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg | Placebo
Number analyzed (Participants) | 45 | 23 | 21 | 51
mm | 0.584 (2.344) | 1.140 (2.986) | 0.304 (2.109) | 0.393 (1.586)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) up to 2 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = 0.28, 95% CI 2-sided [-0.58 to 1.14]
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521) up to 1 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = 0.82, 95% CI 2-sided [-0.23 to 1.87]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -0.03, 95% CI 2-sided [-1.11 to 1.06]

10. Secondary Outcome: Systolic Pulmonary Arterial Pressure (PAPsyst) - Change From Baseline to Week 16
Description: Systolic pulmonary arterial pressure (PAPsyst) is a directly measured hemodynamic parameter acquired during a right heart catheterization.
Time Frame: Baseline and visit 6 (16 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2 mg | Riociguat (Adempas, BAY63-2521) up to 1 mg | Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg | Placebo
Number analyzed (Participants) | 54 | 28 | 22 | 55
mmHg | -7.69 (14.251) | -2.89 (12.333) | -5.86 (11.589) | -4.49 (13.717)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) up to 2 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -3.84, 95% CI 2-sided [-8.76 to 1.09]
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521) up to 1 mg vs Placebo; Test type: Superiority or Other; LS-MEANs Difference = -0.02, 95% CI 2-sided [-6.05 to 6.01]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -2.43, 95% CI 2-sided [-8.93 to 4.06]

11. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF) - Change From Baseline to Week 16
Description: The left ventricular ejection fraction work index (LVEF) is a calculated echocardiography parameter. LVEF is derived from the directly measured parameters left ventricular end-diastolic volume (LVEDV) and left ventricular end-systolic volume (LVESV). These 2 parameters are acquired during a non-invasive echocardiography examination. Formula: LEVF = 100*(LVEDV - LVESV)/LVEDV
Time Frame: Baseline and visit 6 (16 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2 mg | Riociguat (Adempas, BAY63-2521) up to 1 mg | Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg | Placebo
Number analyzed (Participants) | 52 | 27 | 22 | 51
Percentage | 6.599 (43.187) | 12.659 (41.769) | 5.529 (48.322) | 11.121 (42.989)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) up to 2 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = 0.51, 95% CI 2-sided [-0.21 to 1.24]
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521) up to 1 mg vs Placebo; Test type: Superiority or Other; LS_MEANS Difference = 0.81, 95% CI 2-sided [-0.07 to 1.69]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = 0.20, 95% CI 2-sided [-0.74 to 1.15]

12. Secondary Outcome: Left Ventricular End-systolic Volume (LVESV) - Change From Baseline to Week 16
Description: Left ventricular end-systolic volume (LVESV) is a measured echocardiography parameter. It is acquired during a non-invasive echocardiography examination.
Time Frame: Baseline and visit 6 (16 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2 mg | Riociguat (Adempas, BAY63-2521) up to 1 mg | Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg | Placebo
Number analyzed (Participants) | 52 | 27 | 22 | 51
mL | 1.805 (31.735) | 6.415 (28.832) | 1.507 (34.033) | 7.295 (32.311)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) up to 2 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -5.06, 95% CI 2-sided [-17.33 to 7.22]
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521) up to 1 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = 0.28, 95% CI 2-sided [-14.55 to 15.11]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -5.18, 95% CI 2-sided [-21.05 to 10.69]

13. Secondary Outcome: Left Ventricular End-diastolic Volume (LVEDV) - Change From Baseline to Week 16
Description: Left ventricular end-diastolic volume (LVEDV) is a measured echocardiography parameter. It is acquired during a non-invasive echocardiography examination.
Time Frame: Baseline and visit 6 (16 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2 mg | Riociguat (Adempas, BAY63-2521) up to 1 mg | Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg | Placebo
Number analyzed (Participants) | 52 | 27 | 22 | 51
mL | 6.599 (43.187) | 12.659 (41.769) | 5.529 (48.322) | 11.121 (42.989)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) up to 2 mg vs Placebo; Test type: Superiority or Other; LS_MEANS Difference = -4.27, 95% CI 2-sided [-21.13 to 12.60]
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521) up to 1 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = 2.78, 95% CI 2-sided [-17.59 to 23.16]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -4.61, 95% CI 2-sided [-26.43 to 17.20]

14. Secondary Outcome: E-wave Deceleration Time - Change From Baseline to Week 16
Description: E-wave deceleration time is a measured echocardiography parameter. It is acquired during a non-invasive echocardiography examination.
Time Frame: Baseline and visit 6 (16 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2 mg | Riociguat (Adempas, BAY63-2521) up to 1 mg | Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg | Placebo
Number analyzed (Participants) | 49 | 22 | 21 | 53
msec | 2.857 (31.470) | -0.636 (38.138) | 8.000 (39.542) | -1.208 (43.937)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) up to 2 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = 5.29, 95% CI 2-sided [-7.38 to 17.95]
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521) up to 1 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = 6.47, 95% CI 2-sided [-9.79 to 22.73]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = 10.35, 95% CI 2-sided [-6.14 to 26.84]

15. Secondary Outcome: Ratio of Mitral Peak Velocity of Early Filling to Mitral Peak Velocity of Late Filling (E/A) - Change From Baseline to Week 16
Description: E/A ratio is a measured echocardiography parameter and describes the ratio of mitral peak velocity of early filling to mitral peak velocity of late filling. It is acquired during a non-invasive echocardiography examination.
Time Frame: Baseline and visit 6 (16 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: E/A ratio
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2 mg | Riociguat (Adempas, BAY63-2521) up to 1 mg | Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg | Placebo
Number analyzed (Participants) | 44 | 20 | 20 | 48
E/A ratio | -0.247 (0.957) | 0.141 (1.261) | -0.063 (0.884) | -0.175 (1.079)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) up to 2 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -0.15, 95% CI 2-sided [-0.55 to 0.24]
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521) up to 1 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = 0.17, 95% CI 2-sided [-0.34 to 0.67]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = 0.06, 95% CI 2-sided [-0.45 to 0.56]

16. Secondary Outcome: 6-minute Walking Distance (6MWD) - Change From Baseline to Week 16
Description: 6-minute walking distance (6MWD) is a measure for the objective evaluation of a patient's functional exercise capacity.
Time Frame: Baseline and visit 6 (16 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2 mg | Riociguat (Adempas, BAY63-2521) up to 1 mg | Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg | Placebo
Number analyzed (Participants) | 54 | 28 | 22 | 55
m | 31.425 (83.386) | 25.379 (84.244) | -2.784 (90.324) | 17.857 (80.851)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) up to 2 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = 10.17, 95% CI 2-sided [-18.48 to 38.81]
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521) up to 1 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = 7.92, 95% CI 2-sided [-26.76 to 42.59]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -6.15, 95% CI 2-sided [-44.08 to 31.78]

17. Secondary Outcome: WHO (World Health Organization) Functional Class - Change From Baseline to Week 16
Description: The WHO functional assessment of pulmonary arterial hypertension ranged from functional class I (Patients with PH but without resulting limitation of physical activity) to class IV (Patients with PH with inability to carry out any physical activity without symptoms. These patients manifest signs of right-heart failure.). Changes to a lower WHO functional class resemble improvement, changes to a higher functional class resemble deterioration of PAH.
Time Frame: Baseline and visit 6 (16 weeks)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2 mg | Riociguat (Adempas, BAY63-2521) up to 1 mg | Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg | Placebo
Number analyzed (Participants) | 54 | 28 | 22 | 56
Percentage of participants
  -1 | 20.4 | 21.4 | 22.7 | 19.6
  0 | 74.1 | 75 | 68.2 | 71.4
  1 | 5.6 | 3.6 | 9.1 | 8.9

18. Secondary Outcome: Percentage of Participants With Clinical Worsening
Description: The combined endpoint "time to clinical worsening", made up of the following components, defined by the first occurrence: all cause mortality, including cardiovascular mortality; first hospitalization for a cardiovascular event, including heart failure, acute myocardial infarction, stroke or ventricular arrhythmia; upgrade of the HTx (heart transplantation) status to next higher level; need for IV diuretics; persistent worsening of WHO functional class due to deterioration of PH or cardiac function.
Time Frame: At visit 6 (16 weeks)
Population: Intent to Treat (ITT) - a randomized participant was valid for ITT analyses if at least one dose of study medication was administered. Only participants with a baseline and at least one post-baseline measurement were included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2 mg | Riociguat (Adempas, BAY63-2521) up to 1 mg | Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg | Placebo
Number analyzed (Participants) | 67 | 33 | 32 | 69
Percentage of participants | 23.9 | 15.1 | 15.6 | 21.7
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) up to 2 mg vs Placebo; Test type: Superiority or Other; Risk Difference (RD) = 0.62, 95% CI 2-sided [-13.36 to 14.61]
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521) up to 1 mg vs Placebo; Test type: Superiority or Other; Risk Difference (RD) = -9.46, 95% CI 2-sided [-24.32 to 5.39]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg vs Placebo; Test type: Superiority or Other; Risk Difference (RD) = -6.07, 95% CI 2-sided [-22.26 to 10.13]

19. Secondary Outcome: Borg CR 10 Scale - Change From Baseline to Week 16
Description: The Borg CR10 Scale is a patient reported outcome measure used in clinical diagnosis of e.g. breathlessness and dyspnea. It documents the patient's exertion during a physical test. Low values indicate low levels of exertion, high values indicate more intense exertion reported by the patient. The score ranges from 0 ("Nothing at all") to 10 ("Extremely strong - Maximal").
Time Frame: Baseline and visit 6 (16 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2 mg | Riociguat (Adempas, BAY63-2521) up to 1 mg | Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg | Placebo
Number analyzed (Participants) | 54 | 28 | 22 | 55
Scores on a scale | 0.269 (1.900) | -0.804 (2.319) | -0.682 (1.516) | 0.187 (2.640)

20. Secondary Outcome: EQ-5D Utility Score - Change From Baseline to Week 16
Description: EQ-5D utility score is a Quality-of-Life patient reported outcome measure. An increase in the utility score represents an improvement in quality of life. The score ranges from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: Baseline and visit 6 (16 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2 mg | Riociguat (Adempas, BAY63-2521) up to 1 mg | Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg | Placebo
Number analyzed (Participants) | 54 | 28 | 22 | 56
Scores on a scale | 0.073 (0.211) | 0.016 (0.242) | 0.004 (0.166) | 0.018 (0.201)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) up to 2 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = 0.03, 95% CI 2-sided [-0.04 to 0.10]
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521) up to 1 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = 0.01, 95% CI 2-sided [-0.07 to 0.09]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = 0.02, 95% CI 2-sided [-0.07 to 0.11]

21. Secondary Outcome: Minnesota Living With Heart Failure Questionnaire (MLHF) Score - Change From Baseline to Week 16
Description: The self-reported Minnesota Living with Heart Failure questionnaire (MLHF) is designed to measure the effects of PH and PH-specific treatments on an individual's quality of life. The MLHF total score can range from 0 (best) to 105 (worst).
Time Frame: Baseline and visit 6 (16 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2 mg | Riociguat (Adempas, BAY63-2521) up to 1 mg | Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg | Placebo
Number analyzed (Participants) | 54 | 28 | 22 | 55
Scores on a scale | -10.789 (22.232) | -5.132 (14.111) | -7.595 (18.651) | 0.211 (15.964)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) up to 2 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -6.80, 95% CI 2-sided [-12.81 to -0.78]
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521) up to 1 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -6.81, 95% CI 2-sided [-13.96 to 0.35]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -7.50, 95% CI 2-sided [-15.29 to 0.28]

22. Secondary Outcome: Cystatin C - Change From Baseline to Week 16
Description: Cystatin C is a biomarker for predicting new onset or deteriorating cardiovascular disease.
Time Frame: Baseline and visit 6 (16 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2 mg | Riociguat (Adempas, BAY63-2521) up to 1 mg | Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg | Placebo
Number analyzed (Participants) | 45 | 26 | 17 | 44
ng/mL | 39.3 (232.7) | 11.2 (218.5) | 71.2 (140.8) | 58.6 (242.9)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) up to 2 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -24.62, 95% CI 2-sided [-117.58 to 68.33]
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521) up to 1 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -53.29, 95% CI 2-sided [-162.46 to 55.88]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -8.36, 95% CI 2-sided [-135.78 to 119.06]

23. Secondary Outcome: N-terminal Pro-brain Natriuretic Peptide (NT-pro BNP) - Change From Baseline to Week 16
Description: N-terminal pro-brain natriuretic peptide (NT-pro BNP) levels in the blood are used for screening, diagnosis of acute congestive heart failure (CHF) and may be useful to establish prognosis in heart failure.
Time Frame: Baseline and visit 6 (16 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2 mg | Riociguat (Adempas, BAY63-2521) up to 1 mg | Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg | Placebo
Number analyzed (Participants) | 50 | 28 | 21 | 54
pg/mL | -168.42 (1585.28) | -213.48 (1204.24) | -215.71 (769.16) | 171.51 (2123.55)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) up to 2 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -407.34, 95% CI 2-sided [-1055.23 to 240.54]
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521) up to 1 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -447.26, 95% CI 2-sided [-1212.74 to 318.22]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -517.48, 95% CI 2-sided [-1369.48 to 334.53]

24. Secondary Outcome: Troponin T - Change From Baseline to Week 16
Description: Troponin T is a cardiac-specific protein which is released from damaged or injured heart muscle cells.
Time Frame: Baseline and visit 6 (16 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2 mg | Riociguat (Adempas, BAY63-2521) up to 1 mg | Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg | Placebo
Number analyzed (Participants) | 34 | 24 | 15 | 44
µg/L | 0.005 (0.027) | -0.008 (0.042) | -0.001 (0.006) | 0.003 (0.015)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) up to 2 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = 0.00, 95% CI 2-sided [-0.01 to 0.01]
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521) up to 1 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -0.01, 95% CI 2-sided [-0.02 to 0.00]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -0.01, 95% CI 2-sided [-0.02 to 0.01]

25. Secondary Outcome: Asymmetric Dimethylarginine (ADMA) - Change From Baseline to Week 16
Description: Asymmetric dimethylarginine (ADMA) is an endogenous inhibitor of nitric oxides. Recent clinical studies have indicated that ADMA may have diagnostic relevance as a novel cardiovascular risk marker.
Time Frame: Baseline and visit 6 (16 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2 mg | Riociguat (Adempas, BAY63-2521) up to 1 mg | Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg | Placebo
Number analyzed (Participants) | 49 | 25 | 19 | 51
µmol/L | 0.020 (0.115) | 0.026 (0.118) | 0.006 (0.098) | 0.020 (0.090)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) up to 2 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -0.00, 95% CI 2-sided [-0.04 to 0.03]
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521) up to 1 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = 0.00, 95% CI 2-sided [-0.04 to 0.05]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -0.02, 95% CI 2-sided [-0.07 to 0.03]

26. Secondary Outcome: Osteopontin - Change From Baseline to Week 16
Description: Osteopontin is a cytokine-like pro-fibrotic mediator, which is expressed in cardiovascular tissues. Its expression is induced by increased pressure and volume load in the myocardium, kidney and lung. Therefore, osteopontin may be used as a prognostic marker in patients with cardiovascular diseases.
Time Frame: Baseline and visit 6 (16 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2 mg | Riociguat (Adempas, BAY63-2521) up to 1 mg | Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg | Placebo
Number analyzed (Participants) | 50 | 27 | 18 | 51
µg/mL | -13.400 (44.931) | -0.852 (22.396) | -2.722 (29.379) | -4.588 (77.576)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) up to 2 mg vs Placebo; Test type: Superiority or Other; LS-MEANSA Difference = -14.13, 95% CI 2-sided [-30.79 to 2.53]
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521) up to 1 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -12.73, 95% CI 2-sided [-32.89 to 7.43]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg vs Placebo; Test type: Superiority or Other; LS-MEANS Difference = -18.27, 95% CI 2-sided [-41.53 to 5.00]

ADVERSE EVENTS:
Time Frame: All Adverse Events occurring between the subject has signed the informed consent and 30 days after the definite stop of study medication (over a period approximately 25 months) were reported.
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2 mg | Riociguat (Adempas, BAY63-2521) up to 1 mg | Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 23/67 | 7/33 | 7/32 | 18/69
Other Adverse Events (participants affected / at risk) | 57/67 | 28/33 | 25/32 | 49/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riociguat (Adempas, BAY63-2521) up to 2 mg (N=67) | Riociguat (Adempas, BAY63-2521) up to 1 mg (N=33) | Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg (N=32) | Placebo (N=69)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 7 (8) | 3 (4) | 1 (1) | 3 (3)
Cardiac failure acute (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0) | 3 (4)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cyst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hernia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Medical device complication (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device malfunction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device dislocation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperphagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Critical illness polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heart transplant (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac pacemaker replacement (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Implantable defibrillator insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Implantable defibrillator replacement (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haemodynamic instability (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riociguat (Adempas, BAY63-2521) up to 2 mg (N=67) | Riociguat (Adempas, BAY63-2521) up to 1 mg (N=33) | Riociguat (Adempas, BAY63-2521) Fixed 0.5 mg (N=32) | Placebo (N=69)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 4 (4) | 0 (0) | 2 (3)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 6 (7) | 0 (0) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 4 (4) | 0 (0) | 1 (2) | 4 (4)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Pulmonary valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 12 (14) | 5 (11) | 0 (0) | 5 (7)
Dyspepsia (Gastrointestinal disorders) | 6 (8) | 6 (8) | 2 (4) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperchlorhydria (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (11) | 2 (2) | 2 (2) | 5 (7)
Vomiting (Gastrointestinal disorders) | 5 (5) | 2 (2) | 0 (0) | 4 (6)
Chest discomfort (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 2 (3) | 2 (4)
Fatigue (General disorders) | 4 (6) | 0 (0) | 3 (3) | 3 (4)
Oedema peripheral (General disorders) | 5 (6) | 4 (4) | 4 (5) | 5 (6)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 0 (0) | 4 (4)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) | 2 (2)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 3 (3) | 2 (3) | 4 (4)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 7 (7)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 8 (9)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Blood uric acid increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Heart rate decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
International normalised ratio abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 2 (2) | 4 (4) | 1 (1) | 1 (1)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary arterial wedge pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Glutamate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Electrocardiogram repolarisation abnormality (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Occult blood positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (4) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 1 (1) | 3 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appetite disorder (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (2) | 0 (0) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (2) | 1 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (5) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Bone swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 11 (13) | 4 (5) | 5 (7) | 7 (8)
Dizziness postural (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 10 (11) | 4 (4) | 1 (1) | 7 (8)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Orthostatic intolerance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Erection increased (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 4 (4) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (5) | 3 (4) | 9 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Arteriosclerosis Moenckeberg-type (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Haematoma (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 8 (8) | 5 (7) | 3 (5) | 3 (5)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Venous insufficiency (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Subjects had advanced disease and were heavily pretreated. Baseline values were not comparable between treatment groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigative Site, Institution and/or Principal Investigator shall furnish the Sponsor with a copy of any proposed publication of material at least sixty (60) days in advance of the date of submission for publication or presentation.